CLINICAL TRIAL: NCT00837551
Title: A Randomized, Double-Blinded, Vehicle-Controlled Phase IIa Study to Evaluate Topically Applied WBI-1001 Cream in Patients With Atopic Dermatitis.
Brief Title: Phase IIa Study of WBI-1001 Cream for Atopic Dermatitis
Acronym: WBI-1001-201
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Welichem Biotech Inc. (Industry)
Responsible Party: Robert Bissonnette, Innovaderm Reseaerch Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WBI-1001-201: Control # 119727
Record Dates: First submitted 2009-02-03; First posted 2009-02-05 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Dermatitis, Atopic
Keywords: Non-steroid; Small molecule; Topical cream; Inflammatory disease; Skin
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tapinarof

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 Placebo cream (Placebo Comparator): 0% cream 12 patients
  Interventions: Drug: WBI-1001
- 2. Cream (Active Comparator): 0.5% WBI-1001 cream 12 patients
  Interventions: Drug: WBI-1001
- 3. Cream (Active Comparator): 1.0% WBI-1001 cream 12 patients
  Interventions: Drug: WBI-1001

INTERVENTIONS:
Drug: WBI-1001 — Doses of 0,0.5% and 1.0% cream. Topical cream application. Twice daily for 28 days. Duration of treatment: 28 days with one week follow-up.

SUMMARY:
WBI-1001 is a synthetic,new, non-steroid, small molecule being developed as a candidate drug for the topical, cream treatment of inflammatory skin diseases. As such, it affects T-cells through inhibition of T-cell activities including their infiltration processes, and it shows direct anti-inflammatory manifestation in the mouse edema model. This was a 28 day study (plus one follow-up week) on patients with Atopic Dermatitis, and 36 patients were treated randomly, BID with either 0.5%, 1.0% or placebo. Blood samples were taken weekly for PK analysis.

DETAILED DESCRIPTION:
A double-blind, single-centered, vehicle-controlled, randomized Phase IIa study of WBI-1001 on patients with mild to moderate Atopic Dermatitis (AD). All body areas were treatable except face, scalp, groin and genital areas. Cream applied BID between 6.00 and 10.00am and 7.00 and 10.00pm daily for 4 weeks. Blood draws for PK analysis were taken weekly at the study centre prior to the morning cream application. Patients returned to the study centre approximately one week later for a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* AD diagnosis (based on Hanifin's criteria) presenting a minimum of 1% and a maximum of 10% body surface area (BSA) excluding face, groin, scalp and genital areas.
* Disease severity index (EASI) of less than 12, Investigator's Global Assessment (IGA) of 2-3 at Day 0.
* In good general health and free of any condition that might impair evaluation of AD.
* Women of child bearing potential (WOCBP) had to have a negative a negative serum human-beta chorionic gonadotropin pregnancy test before randomization.

WOCBP had to abstain from sex or they and their partners had to use adequate contraceptive precautions for the duration of the study.

* Willing and able to comply with the protocol and attend all study visits.
* Provide a written informed consent form prior to initiation of study procedures.

Exclusion Criteria:

* Had spontaneously improving or rapidly deteriorating AD.
* Had AD lesions on only hands and/or feet.
* Had skin diseases other than AD.
* Had active allergic contact dermatitis or other non-atopic forms of dermatitis.
* Had other concomitant medical condition that could put the patient at risk during the study.
* Had a history of neurological/psychiatric disorders that could interfere with the patient's participation.
* Had systemic immunomodulatory therapies within 12 weeks prior to the baseline visit.
* Had prolonged exposure to natural or artificial ultraviolet radiation within 4 weeks of baseline visit.
* Had phototherapy (including laser), photo-chemotherapy or systemic AD therapy within 4 weeks prior to baseline visit.
* Had topical AD therapies in the areas to be treated within 2 weeks prior to the baseline visit.
* Had alcohol abuse in the last 2 years.
* Had allergic history to any non-medical ingredients of the study cream.
* Were treated with an investigational drug within 1 month of Day 0 or were currently participating in another trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To evaluate skin lesion condition as a measure of safety and tolerability of WBI-1001 treated AD patients. | 0, 7, 14, 21, 28 and 35 days

SECONDARY OUTCOMES:
Assess systemic exposure of WBI-1001 treated AD patients by measuring plasma PK. | 0, 7, 14, 21 and 28 days
Explore efficacy of topically applied WBI-1001 cream in patients with AD. | 0, 7, 14, 21, 28 and 35 days.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research Inc.
Locations (1):
- Innovaderm Research Inc.,, Montreal, Quebec, Canada